CLINICAL TRIAL: NCT06377995
Title: Effectiveness of an Intervention Plan Targeting the Diaphragm in Young Adults With Chronic Non-specific Neck Pain: Randomised Clinical Trial
Brief Title: Effectiveness of an Intervention Plan Aimed at the Diaphragm in Chronic Non-specific Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Teacher, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OST1_013
Record Dates: First submitted 2024-04-05; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Neck Pain
Keywords: Neck pain; Diaphragm; Cervical spine; Young adult; Osteopathy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: Control group (Placebo Comparator): Participants in the control group first rate their pain from 0 to 10 using the Numerical Pain Scale, at rest and at the end of the available range of lateral flexion and rotation. The amplitude of these movements is then assessed using a Goniometer Pro© (G-pro©). This assessment takes 10 minutes.
  After the initial assessment, the researcher performs the placebo technique, which lasts 12 minutes. Finally, the initial assessment is carried out again.
  Interventions: Other: Placebo technique
- Experimental: Diaphragm protocol (Experimental): Participants in the experimental group first rate their pain from 0 to 10 using the Numerical Pain Scale, at rest and at the end of the available range of lateral flexion and rotation. The amplitude of these movements is then assessed using a Goniometer Pro© (G-pro©). This assessment takes 10 minutes.
  After the initial assessment, the researcher performs the diaphragm stretching, neuromuscular and phrenic centre inhibition technique; this treatment protocol lasts 12 minutes.
  Finally, the initial assessment is carried out again
  Interventions: Other: Diaphragm protocol

INTERVENTIONS:
Other: Placebo technique — The patient is in a supine position with a 90° knees flexion. The osteopath lies cephalad to the patient and places their hands on their shoulders.
  Arms: Placebo Comparator: Control group
Other: Diaphragm protocol — The patient is in a supine position with a 90° knees flexion.To stretch the diaphragm, the osteopath stands at the head of the bed and places his hands on the lower edge of the ribcage and accompanies the lifting of the ribs during inhalation and maintains it during deep exhalation for up to 2 sets of 10 deep breaths separated by 1 minute. For the neuromuscular technique, the osteopath is positioned contralateral to the side to be treated and slides with the thumb under the lower part of the thorax, applying a force in the opposite direction.To inhibit the phrenic centre, the osteopath places one hand on the sternum in a caudal direction and the other in the projection of the phrenic centre in a cephalic direction.The participant inhales deeply and the osteopath presses in both directions during the expiratory phase for 10 respiratory cycles.
  Arms: Experimental: Diaphragm protocol

SUMMARY:
The aim of this study is to analyse the effectiveness of an intervention plan targeting the diaphragm, namely stretching technique, neuromuscular diaphragm and phrenic centre inhibition, in the treatment of chronic non-specific neck pain.

DETAILED DESCRIPTION:
Chronic neck pain is defined as pain and discomfort between the superior nuchal line and the spinous process of the first thoracic vertebra, which may radiate to the scapula, anterior chest wall, skull or upper limbs. It is classified as chronic if the pain persists for more than 12 weeks. Associated symptoms include headache, dizziness and pain or paresthesia in the upper limbs. These symptoms interfere with daily life and have a negative impact on physical and mental health.

The aetiology of this pathology is multifactorial and the triggering factors may vary due to the close relationship that the cervical spine has with other structures, namely the diaphragm muscle.

Our aim is to verify the effectiveness of an osteopathic treatment protocol targeting the diaphragm in chronic non-specific neck pain in young adults. Specifically, to analyse whether the mechanical, fascial and neural pathways established by the defined manual techniques, namely stretching techniques, neuromuscular inhibition of the diaphragm and the phrenic centre, have any effect on active movements (rotations and inclinations) and chronic neck pain.

This study will analyse the effects of diaphragmatic techniques on the following variables: Numerical Pain Scale and Goniometer Pro© (G-pro©).

ELIGIBILITY:
Inclusion Criteria:

* Present a negative Jackson test;
* Have a body mass index (BMI) of 20-29.9 kg/m2;
* Suffer from chronic non-specific neck pain for 3 months or more.

Exclusion Criteria:

* Have a history of cervical spine surgery, as well as any trauma or fracture of the cervical spine, clavicle, scapula and ribs;
* Have specific neck pain due to degenerative diseases (disc prolapse, scoliosis);
* Having a congenital cervical deformity, such as torticollis;
* Being pregnant;
* Having rheumatic, oncological or respiratory pathologies;
* Have liver or gallbladder pathologies;
* Receiving physiotherapy, osteopathy, acupuncture or massage treatment for neck pain 3 months before and during participation in the study;
* Taking analgesics, anti-inflammatories or muscle relaxants 5 days prior to the intervention.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the intensity of pain in the cervical spine after applying the diaphragm intervention plan | 12 minutes after the intervention
  The questionnaire of Numerical Pain Scale (NPS) will be the instrument used to access the volunteer's pain, which consists of a numerical scale from 0 to 10, in which 0 is absence of pain and 10 is maximal pain. This questionnaire is carried out at rest and at the end of the available range of lateral inclinations and rotations of the cervical spine, which are the most painful movements in this pathology.
Changes in range of motion after applying the diaphragm targeted protocol | 12 minutes after the intervention
  The range of motion of the cervical spine, rotations and lateral inclinations will be measured using the Goniometer Pro© (G-pro©) to compare the pre- and post-intervention samples.
  NPS questionnaire data will be collected from the subject's report and recorded in an Excel spreadsheet with the appropriate identification code.
  The range of motion data will be collected by the assessor and recorded in an Excel spreadsheet with the appropriate identification code.

SECONDARY OUTCOMES:
Changes in pain level one week after the intervention | One week after the intervention.
  One week later, the volunteers will take the Numerical Pain Scale (NPS) questionnaire again to access the volunteers pain, which consists of a numerical scale from 0 to 10, where 0 is no pain and 10 is maximum pain. This questionnaire is carried out at rest and at the end of the available range of lateral inclinations and rotations of the cervical spine, which are the most painful movements in this pathology.
Changes in range of motion one week later | One week after the intervention.
  The range of motion of the rotation and lateral tilt of the cervical spine is measured again using a Goniometer Pro© (G-pro©).
  Data from the NPS questionnaire will be collected from the patient report and recorded in an Excel document with the corresponding identification code.
  The range of motion data is collected by the assessor and recorded in an Excel spreadsheet with the appropriate identification code.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior da Saúde do Porto
Locations (1):
- Escola Superior de Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Ahmad, A., Kamel, K. M., & Mohammed, R. G. (2020). Effect of forward head posture on diaphragmatic excursion in subjects with chronic neck pain. a case-control study. Physiotherapy Quarterly, 28(3), 9-13. https://doi.org/10.5114/pq.2020.95769
- [Background] Chaitow, L., & Delany, J. (2008). Clinical application of neuromuscular techniques. Volume 1, The upper body. Churchill Livingstone Elsevier.
- [Background] Haghighat F, Moradi R, Rezaie M, Yarahmadi N, Ghaffarnejad F. Added value of diaphragm myofascial release on forward head posture and chest expansion in women with symptomatic forward head posture: A randomized controlled trial. J Bodyw Mov Ther. 2025 Dec;45:645-651. doi: 10.1016/j.jbmt.2025.07.015. Epub 2025 Aug 8. PMID 41316631
- [Background] Haller H, Lauche R, Cramer H, Rampp T, Saha FJ, Ostermann T, Dobos G. Craniosacral Therapy for the Treatment of Chronic Neck Pain: A Randomized Sham-controlled Trial. Clin J Pain. 2016 May;32(5):441-9. doi: 10.1097/AJP.0000000000000290. PMID 26340656
- [Background] Mármol, M. (2023). Efectos de la maniobra de inhibición fascial del diafragma sobre la columna cervical en pacientes con cervicalgia inespecífica. Revista de Investigación Osteopática, 3 (1), 22-28.
- [Background] Silva ACO, Biasotto-Gonzalez DA, Oliveira FHM, Andrade AO, Gomes CAFP, Lanza FC, Amorim CF, Politti F. Effect of Osteopathic Visceral Manipulation on Pain, Cervical Range of Motion, and Upper Trapezius Muscle Activity in Patients with Chronic Nonspecific Neck Pain and Functional Dyspepsia: A Randomized, Double-Blind, Placebo-Controlled Pilot Study. Evid Based Complement Alternat Med. 2018 Nov 11;2018:4929271. doi: 10.1155/2018/4929271. eCollection 2018. PMID 30534176
- [Background] Simoni G, Bozzolan M, Bonnini S, Grassi A, Zucchini A, Mazzanti C, Oliva D, Caterino F, Gallo A, Da Roit M. Effectiveness of standard cervical physiotherapy plus diaphragm manual therapy on pain in patients with chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:481-491. doi: 10.1016/j.jbmt.2020.12.032. Epub 2021 Feb 16. PMID 33992285
- [Background] Tatsios PI, Grammatopoulou E, Dimitriadis Z, Papandreou M, Paraskevopoulos E, Spanos S, Karakasidou P, Koumantakis GA. The Effectiveness of Spinal, Diaphragmatic, and Specific Stabilization Exercise Manual Therapy and Respiratory-Related Interventions in Patients with Chronic Nonspecific Neck Pain: Systematic Review and Meta-Analysis. Diagnostics (Basel). 2022 Jun 30;12(7):1598. doi: 10.3390/diagnostics12071598. PMID 35885502
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Rosas S, Paco M, Lemos C, Pinho T. Comparison between the Visual Analog Scale and the Numerical Rating Scale in the perception of esthetics and pain. Int Orthod. 2017 Dec;15(4):543-560. doi: 10.1016/j.ortho.2017.09.027. Epub 2017 Nov 13. PMID 29146313
- [Background] Pourahmadi MR, Bagheri R, Taghipour M, Takamjani IE, Sarrafzadeh J, Mohseni-Bandpei MA. A new iPhone application for measuring active craniocervical range of motion in patients with non-specific neck pain: a reliability and validity study. Spine J. 2018 Mar;18(3):447-457. doi: 10.1016/j.spinee.2017.08.229. Epub 2017 Sep 7. PMID 28890223